CLINICAL TRIAL: NCT04679818
Title: Postoperative Consequences of Intraoperative NOL Titration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-1646
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Adverse Effect
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- PMD-200 NOL group (Active Comparator): Clinicians will titrate fentanyl to keep PMD-200 (Pain Monitoring Device) Nociception level (NOL) under 25 - always using good clinical judgement for individual patients
  Interventions: Device: PMD-200 Nol-guided opioid administration
- Control Group (Active Comparator): Clinicians will be blinded to PMD-200 Nociception level (NOL) monitoring and use clinical judgement to determine how much fentanyl should be given, and when.
  Interventions: Drug: Routine opioid management

INTERVENTIONS:
Drug: Routine opioid management — Clinical judgement will be according to their standard practice and may include interpretation of blood pressure, heart rate, diaphoresis, tearing, and pupil size. Boluses of fentanyl 1 µg/kg actual body weight (ABW), up to a maximum dose of 100 µg per bolus, can be given per clinical judgement.
  Other Names: Fentanyl
  Arms: Control Group
Device: PMD-200 Nol-guided opioid administration — PMD-200 Nociception level (NOL) values exceeding 25 for more than 30 seconds will typically be treated with boluses of fentanyl 1µg/kg ABW, up to a maximum of 100 µg per boluses, 5-minute intervals. Towards the end of the surgery (approximately 30-45 minutes before end of surgery, based on clinical judgment), the boluses of fentanyl will be reduced to 0.5 µg/kg ABW, up to a maximum of 50 µg per boluses, 5 minutes intervals. The target of a PMD-200 NOL score below 25 will be maintained until surgery ends
  Other Names: PMD-200 NOL
  Arms: PMD-200 NOL group

SUMMARY:
To demonstrate that intraoperative NOL-guided titration of fentanyl improves initial recovery characteristics.

DETAILED DESCRIPTION:
Previous work has shown that NOL (Nociception Level) accurately quantifies nociception during general anesthesia.6 Presumably, titrating opioids to NOL will therefore provide individual guidance so that patients will be given about the right amount. Patient given the right amount will presumably awaken quickly when anesthesia is done, and have good initial pain control in the PACU (Post-Anesthesia Care Unit). To the extent that NOL titration facilitates optimal opioid dosing, patients are likely to have better PACU experiences - which would be an important outcome that clinicians and regulators are likely to take seriously.

ELIGIBILITY:
Inclusion Criteria:

* Adults having major non-cardiac surgery expected to last ≥2 hours
* American Society of Anesthesiologists physical status 1-3
* Age 21-85 years old
* Planned endotracheal intubation

Exclusion Criteria:

* Planned neuraxial or regional block
* Clinician preference for an opioid other than, or in addition to, fentanyl
* Non-sinus heart
* Neurologic condition that, in the opinion of the investigators, may preclude accurate assessment of postoperative pain and nausea
* Lack of English language fluency
* Routine user of psychoactive drugs other than opioids
* Contraindication to sevoflurane, fentanyl, morphine, or ondansetron.
* Intracranial surgery.
* BMI > 40

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Ruetzler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ruetzler K, Montalvo M, Bakal O, Essber H, Rossler J, Mascha EJ, Han Y, Ramachandran M, Keebler A, Turan A, Sessler DI. Nociception Level Index-Guided Intraoperative Analgesia for Improved Postoperative Recovery: A Randomized Trial. Anesth Analg. 2023 Apr 1;136(4):761-771. doi: 10.1213/ANE.0000000000006351. Epub 2023 Jan 20. PMID 36727855

RESULTS

PARTICIPANT FLOW:
Groups:
- PMD-200 NOL Group: Clinicians will titrate fentanyl to keep PMD-200 Nociception level (NOL) under 25 - always using good clinical judgement for individual patients
  PMD-200 Nol-guided opioid administration: PMD-200 NOL values exceeding 25 for more than 30 seconds will typically be treated with boluses of fentanyl 1µg/kg actual body weight (ABW), up to a maximum of 100 µg per boluses, 5-minute intervals. Towards the end of the surgery (approximately 30-45 minutes before end of surgery, based on clinical judgment), the boluses of fentanyl will be reduced to 0.5 µg/kg ABW, up to a maximum of 50 µg per boluses, 5 minutes intervals. The target of a PMD-200 NOL score below 25 will be maintained until surgery ends
- Control Group: Clinicians will be blinded to PMD-200 NOL monitoring and use clinical judgement to determine how much fentanyl should be given, and when.
  Routine opioid management: Clinical judgement will be according to their standard practice and may include interpretation of blood pressure, heart rate, diaphoresis, tearing, and pupil size. Boluses of fentanyl 1 µg/kg actual body weight (ABW), up to a maximum dose of 100 µg per bolus, can be given per clinical judgement.
Period: Overall Study
Arm/Group | PMD-200 NOL Group | Control Group
Started | 35 | 37
Completed | 34 | 37
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PMD-200 NOL Group: Clinicians will titrate fentanyl to keep PMD-200 NOL under 25 - always using good clinical judgement for individual patients
  PMD-200 Nol-guided opioid administration: PMD-200 NOL values exceeding 25 for more than 30 seconds will typically be treated with boluses of fentanyl 1µg/kg ABW, up to a maximum of 100 µg per boluses, 5-minute intervals. Towards the end of the surgery (approximately 30-45 minutes before end of surgery, based on clinical judgment), the boluses of fentanyl will be reduced to 0.5 µg/kg ABW, up to a maximum of 50 µg per boluses, 5 minutes intervals. The target of a PMD-200 NOL score below 25 will be maintained until surgery ends
- Total: Total of all reporting groups
Arm/Group | PMD-200 NOL Group | Control Group | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (16) | 54 (15) | 56 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 19 | 18 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 33 | 64
  Other | 4 | 4 | 8
Height [Mean (Standard Deviation); unit: cm] | 171 (11) | 171 (10) | 171 (10)
Weight [Mean (Standard Deviation); unit: kg] | 78 (19) | 82 (23) | 80 (21)
BMI [Mean (Standard Deviation); unit: kg/m2] | 27 (5) | 28 (6) | 28 (6)
Procedure type [Count of Participants; unit: Participants]
  Open | 21 | 15 | 36
  Laparoscopy | 14 | 22 | 36
Surgery type [Count of Participants; unit: Participants]
  Colorectal | 34 | 25 | 59
  Hernia | 1 | 0 | 1
  Other | 0 | 2 | 2
ASA (American Society of Anesthesiologist) physical status [Count of Participants; unit: Participants] — ASA I: A normal healthy patient (better) ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease (worse)
  Participants
    I (healthy) | 0 | 1 | 1
    II (mild systemic disease) | 10 | 8 | 18
    III (severe systemic disease) | 25 | 28 | 53
Preoperative opioid use [Count of Participants; unit: Participants] | 3 | 3 | 6
Preoperative antihypertension medication use [Count of Participants; unit: Participants] | 9 | 15 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores at 10-minute Intervals for the Initial Hour of Recovery
Description: Pain scores are measured using a Verbal Response Scale (VRS) every 10 minutes in the initial hour of recovery. VRS is a scale from 0 to 10 where 0 signifies no pain and 10 signifies the worst pain ever experienced.
Time Frame: At 10-minute intervals during the first 60 minutes after extubation.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
score on a scale
  Time point 1 | 0 [0 to 5.0] | 0 [0 to 4.0]
  Time point 2 | 1.0 [0 to 5.5] | 5.0 [0 to 7.0]
  Time point 3 | 2.5 [0 to 7.0] | 5.0 [2.0 to 7.0]
  Time point 4 | 5.0 [0 to 6.0] | 4.0 [2.0 to 6.0]
  Time point 5 | 4.5 [1.0 to 7.0] | 3.0 [2.0 to 6.0]
  Time point 6 | 4.5 [2.0 to 7.0] | 3.0 [1.0 to 6.0]
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Superiority; p = 0.895, Mixed Models Analysis; Mean Difference (Final Values) = 0.08, 99% CI 2-sided [-1.43 to 1.58]

2. Primary Outcome: Pain Scores at 10-minute Intervals for the Initial 30 Minutes of Recovery
Description: Pain scores are measured using a Verbal Response Scale (VRS) at 10-minute intervals for the initial 30 minutes of recovery. VRS is a scale from 0 to 10 where 0 signifies no pain and 10 signifies the worst pain ever experienced.
Time Frame: At 10-minute intervals during the first 30 minutes after extubation.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
score on a scale
  Time point 1 | 0 [0 to 5.0] | 0 [0 to 4.0]
  Time point 2 | 1.0 [0 to 5.5] | 5.0 [0 to 7.0]
  Time point 3 | 2.5 [0 to 7.0] | 5.0 [2.0 to 7.0]
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Superiority; p = 0.228, Mixed Models Analysis; Mean Difference (Final Values) = -0.84, 99% CI 2-sided [-2.66 to 0.99]

3. Secondary Outcome: Number of Measurements With Pain Score Less Than 5 (vs ≥5) for Initial Hour of Recovery
Description: Binary repeated-measures outcome of pain score will be defined as a pain score less than 5 (vs ≥5). Pain scores will be measured using a Verbal Response Scale (VRS) at 10-minute intervals for the initial hour of recovery. VRS is a scale from 0 to 10 where 0 signifies no pain and 10 signifies the worst pain ever experienced.
Time Frame: At 10-minute intervals during the first 60 minutes after extubation.
Measure: Number; unit: measurements
Units Other Than Participants: Measurements
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
Number analyzed (Measurements) | 196 | 217
measurements | 112 | 130
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Superiority; p = 0.565, generalized linear mixed effects model; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.40 to 1.65]

4. Secondary Outcome: Number of Measurements With Pain Score Less Than 5 (vs ≥5) for the Initial 30 Minutes of Recovery
Description: Binary repeated-measures outcome will be defined as a pain score less than 5 (vs ≥5). Pain scores will be measured using a Verbal Response Scale (VRS) at 10-minute intervals for the 30 minutes of recovery. VRS is a scale from 0 to 10 where 0 signifies no pain and 10 signifies the worst pain ever experienced.
Time Frame: At 10-minute intervals during the first 30 minutes after extubation.
Measure: Number; unit: measurements
Units Other Than Participants: Measurements
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
Number analyzed (Measurements) | 95 | 109
measurements | 63 | 61
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Superiority; p = 0.379, Generalized linear mixed effects model; Risk Ratio (RR) = 1.48, 95% CI 2-sided [0.62 to 3.54]

5. Other Pre Specified Outcome: Number of Analgesic Rescue Boluses
Description: Number of analgesic rescue boluses in the first 60 minutes after extubation.
Time Frame: During the first 60 minutes after extubation.
Measure: Median (Inter-Quartile Range); unit: Number of boluses
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
Number of boluses | 1 [0 to 2] | 2 [0 to 3]
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Superiority; p = 0.039, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.54, 95% CI 2-sided [0.30 to 0.97]

6. Other Pre Specified Outcome: Ramsay Scores During the First 60 Minutes
Description: Ramsay scores will be measured using Ramsay Sedation Scale every 10 minutes in the initial hour of recovery. Ramsay Sedation Scale: 1 = Patient is anxious and agitated or restless, or both; 2 = Patient is co-operative, oriented, and tranquil; 3 = Patient responds to commands only; 4 = Patient exhibits brisk response to light glabellar tap or loud auditory stimulus; 5 = Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus; 6 = Patient exhibits no response. Frequencies for each score were reported.
Time Frame: At 10-minute intervals during the first 60 minutes after extubation.
Measure: Number; unit: Measurements
Units Other Than Participants: Measurements
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
Number analyzed (Measurements) | 203 | 221
Measurements
  1 (Patient is anxious and agitated or restless) | 0 | 1
  2 (Patient is co- operative, oriented, and tranquil) | 92 | 85
  3 (Patient responds to commands only) | 106 | 132
  4 (Patient exhibits brisk response to light glabellar tap or loud auditory stimulus) | 5 | 3
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Non-Inferiority — We tested noninferiority of NOL to routine care on the Ramsey score using an a priori-defined noninferiority delta of 1.2 for the proportional odds ratio; NOL would be deemed noninferior if the upper confidence limit for the odds ratio was <1.2; p = 0.169, proportional odds model; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.35 to 1.82]

7. Other Pre Specified Outcome: Treatment Effect on the Time to Emergence From Anesthesia.
Description: Time to emergence from anesthesia is defined as minutes from discontinuation of sevoflurane anesthesia to extubation
Time Frame: From discontinuation of sevoflurane anesthesia to extubation intraoperatively, assessed up to the timepoint of leaving operation room.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | PMD-200 NOL Group | Control Group
Number analyzed (Participants) | 34 | 37
minutes | 18 [16 to 22] | 20 [18 to 22]
Statistical Analysis 1: Comparison: PMD-200 NOL Group vs Control Group; Test type: Superiority; p = 0.967, Cox proportional hazards regression; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.63 to 1.63]

ADVERSE EVENTS:
Time Frame: From the start of surgery to the initial hour of recovery.
Arm/Group | PMD-200 NOL Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04679818/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT04679818/ICF_003.pdf